CLINICAL TRIAL: NCT06204198
Title: Analysis of Clinicopathological Features and Molecular Typing of Invasive Fibroma of Abdominal Wall and Construction of Recurrence Risk Model
Brief Title: Clinicopathological Features and Molecular Typing of Invasive Fibroma of Abdominal Wall
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Teng Qiong, Resident physician, Shandong Provincial Hospital
Other Study IDs: SWYX:NO.2023-601
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Aggressive Fibromatosis of Abdominal Wall (Disorder)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Surgical retained or paraffin specimens were obtained from patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Aggressive fibromatosis, also known as desmoid fibromatosis or desmoid tumor, is a fibrous tumor that occurs in the fascia, aponeurosis, or deep soft tissue and is formed by excessive proliferation of fibroblasts and myofibroblasts. At present, the disease is considered to be a borderline tumor. Due to the unclear boundary of the tumor, it often grows into the surrounding adjacent tissues, which is difficult to remove completely and easy to relapse. It has been reported that nuclear β-catenin expression and CTNNB1 gene mutation can be used for the differential diagnosis of aggressive fibromatosis from other spindle cell lesions. At present, there is a lack of multicenter retrospective clinical study of this disease, and there is no literature report on the postoperative quality of life of this kind of patients. This study intends to further explore the clinicopathological features, prognosis and molecular typing of abdominal wall aggressive fibroma by retrospective analysis of the case data of multiple hospitals, as well as sequencing analysis of the retained specimens and paraffin specimens from previous operations, to study the high risk factors for recurrence of the disease, and to further comprehensively analyze the impact of abdominal wall aggressive fibroma surgery on the quality of life of patients through follow-up.

DETAILED DESCRIPTION:
The data of all patients with abdominal wall aggressive fibroma were collected through the medical record system of the hospital, and the molecular characteristics of the disease were analyzed by sequencing of the specimens retained by previous surgery or paraffin specimens. The quality of life of patients was investigated by telephone or wechat follow-up to analyze the impact of postoperative disease on the quality of life of patients. As a retrospective and observational study, the data of this study will be statistically summarized according to the following general principles. Categorical data will be summarized descriptively using statistics including frequency n and percentage %, with 95% confidence intervals for overall percentages when necessary, and compared by chi-square or Fisher's exact test. Continuous data will be statistically described as mean ± standard deviation or median (min, Max) and compared by Mann-Whitney (U) test or t-test. The Kaplan-Meier method was used to estimate the survival function for time-to-event data, and survival curves were drawn to estimate the median time and 95% confidence intervals. The differences between groups were compared with the use of the Log-rank test. Cox proportional hazards model was used for univariate and multivariate analysis to screen independent prognostic factors related to recurrence, and the 95% confidence interval (CI) was recorded. All statistical tests were performed with the use of a two-sided 0.05 level. Statistical analysis will be calculated using SPSS 25 statistical analysis software.

ELIGIBILITY:
Inclusion Criteria:

* ① Surgical treatment for "invasive fibroma of abdominal wall"; ② Complete clinical data; ③ Agree to participate in the project.

Exclusion Criteria:

* ① can not cooperate with the project implementation; ② There is cognitive dysfunction; Refuse to participate in research projects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent resection at our hospital for aggressive fibroma in the abdominal wall.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinicopathological features checklist | From September 2023 to September 2024
  Clinicopathological features
Postoperative survival of patients | From September 2023 to September 2024
  Prognosis
Scores of patients' quality of life after surgery | From September 2023 to September 2024
  Patients' quality of life after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yulong Shi, MD, Study Chair — Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China